CLINICAL TRIAL: NCT04474405
Title: An Exploratory Evaluation of the Tau Protein Binding Properties, Whole-Body Biodistribution and Safety of 18F-AV-1451 Injection in Healthy Volunteers and Cognitively Impaired Subjects
Brief Title: Exploratory Evaluation of Flortaucipir Injection in Healthy Volunteers and Cognitively Impaired Subjects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-AV-1451-A01
Record Dates: First submitted 2020-07-08; First posted 2020-07-16 (Actual); Results first posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole; florbetapir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Brain flortaucipir PET scan (Experimental): Subjects receiving a brain PET scan after flortaucipir administration
  Interventions: Drug: Flortaucipir F18; Procedure: Brain PET Scan; Drug: Florbetapir F 18; Procedure: Brain MRI
- Whole body flortaucipir PET scan (Experimental): Subjects receiving a whole body PET scan after flortaucipir administration
  Interventions: Drug: Flortaucipir F18; Procedure: Whole body PET scan
- MRI and Amyloid Extension Cohort (Other): Magnetic resonance imaging (MRI) scans and amyloid scans for subjects previously participating in Study T807000 (NCT01733355)
  Interventions: Procedure: Brain PET Scan; Drug: Florbetapir F 18; Procedure: Brain MRI

INTERVENTIONS:
Drug: Flortaucipir F18 — IV injection, 370 MBq (10 mCi), single dose
  Other Names: 18F-AV-1451; [F-18]T807; LY3191748; Tauvid
  Arms: Brain flortaucipir PET scan; Whole body flortaucipir PET scan
Procedure: Brain PET Scan — positron emission tomography (PET) scan of the brain starting immediately after administration (60 minute dynamic imaging plus 4 frames x 5 minutes at approximately 80 minutes post-dose).
  Arms: Brain flortaucipir PET scan; MRI and Amyloid Extension Cohort
Procedure: Whole body PET scan — positron emission tomography (PET) scan of the body from the vertex of the head to the thighs starting immediately following injection and repeated over 6 hours
  Arms: Whole body flortaucipir PET scan
Drug: Florbetapir F 18 — IV injection, 370 MBq (10 mCi), single dose
  Other Names: Amyvid
  Arms: Brain flortaucipir PET scan; MRI and Amyloid Extension Cohort
Procedure: Brain MRI — Volume-based T1-weighted Magnetic Resonance Imaging (MRI) of the brain
  Arms: Brain flortaucipir PET scan; MRI and Amyloid Extension Cohort

SUMMARY:
This early phase 1 study explored the brain uptake, retention, and safety of flortaucipir and obtained preliminary information regarding dosimetry of flortaucipir.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers had an Mini-Mental State Examination (MMSE) score of ≥ 29;
* MCI due to Alzheimer's disease (AD) consistent with National Institute on Aging (NIA)-Alzheimer's Association working group's on diagnostic guidelines for AD (Alzheimer's Dementia 7:270-9, 2011)
* Possible or probable AD: Met clinical criteria for possible or probable AD based on the NIA-Alzheimer's Association working group's on diagnostic guidelines for AD (Alzheimer's Dementia 7:263-9, 2011)

Exclusion Criteria:

* Current clinically significant psychiatric disease.
* Evidence of structural abnormalities such as major stroke or mass on MRI that would have made a diagnosis of impairment due to AD unlikely or was likely to interfere with interpretation of a PET scan on MRI.
* Claustrophobic or otherwise unable to tolerate the imaging procedure.
* Current clinically significant cardiovascular disease or clinically significant abnormalities on screening electrocardiogram (including, but not limited to, corrected QT interval >450 msec).
* Current clinically significant infectious disease, endocrine or metabolic disease, pulmonary, renal or hepatic impairment, or cancer
* History of alcohol abuse or substance abuse or dependence
* Female subjects of childbearing potential who were not surgically sterile, not refraining from sexual activity or not using reliable methods of contraception.
* Required medications with a narrow therapeutic window
* Received a non-study related radiopharmaceutical imaging or treatment procedure within 7 days prior to imaging session
* Receiving any investigational medications or had participated in a trial with investigational medications within the last 30 days

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-08-16 (Actual); Primary Completion 2013-12-09 (Actual); Study Completion 2013-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Avid Radiopharmaceuticals, Inc.
Locations (2):
- United States (2):
  - WCCT Global, LLC, Cypress, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred between Aug and Dec 2013. Subjects in the MRI and Amyloid Extension cohort received flortaucipir brain PET scans in Study T807000 (NCT01733355)
Pre-assignment Details: Subjects enrolled in the MRI/amyloid extension cohort were to be combined with the Brain PET subgroups for analysis per protocol. MRI allows previously-obtained flortaucipir scan and cognitive data to be combined with the PET scan results from the Brain PET subgroups for analysis.
Groups:
- Brain PET Scan (AD Subjects): Alzheimer's disease (AD) subjects receiving a flortaucipir and florbetapir PET scan
- Brain PET (MCI Subjects): Mild cognitive impairment (MCI) subjects receiving a florbetapir and a flortaucipir PET scan
- Brain PET (YCN Subjects): Young cognitively normal (YCN) subjects receiving florbetapir and a flortaucipir PET scan
- Brain PET (OCN Subjects): Older cognitively normal (OCN) subjects receiving a florbetapir and a flortaucipir PET scan
- Whole Body PET Scan: Subjects receiving a whole body PET scan after flortaucipir administration
- MRI and Amyloid Extension Cohort: Magnetic resonance imaging (MRI) scans and amyloid scans for subjects previously participating in Study T807000. [n=3 AD, n=2 MCI, n=1 OCN]
Period: Overall Study
Arm/Group | Brain PET Scan (AD Subjects) | Brain PET (MCI Subjects) | Brain PET (YCN Subjects) | Brain PET (OCN Subjects) | Whole Body PET Scan | MRI and Amyloid Extension Cohort
Started | 4 | 3 | 5 | 4 | 13 | 7
Flortaucipir PET Scan | 4 | 3 | 4 | 4 | 9 | 0
Florbetapir PET Scan | 4 | 3 | 0 | 4 | 0 | 4
Completed | 4 | 3 | 4 | 4 | 9 | 7
Not Completed | 0 | 0 | 1 | 0 | 4 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Baseline demographics analysis includes subjects receiving a florbetapir or a flortaucipir PET scan in the study.
Groups:
- Brain PET Scan (AD Subjects): AD subjects receiving a flortaucipir and florbetapir PET scan
- Total: Total of all reporting groups
Arm/Group | Brain PET Scan (AD Subjects) | Brain PET (MCI Subjects) | Brain PET (YCN Subjects) | Brain PET (OCN Subjects) | Whole Body PET Scan | MRI and Amyloid Extension Cohort | Total
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 9 | 4 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (7.87) | 78.7 (2.89) | 27.5 (2.08) | 66.3 (0.50) | 56.3 (4.42) | 73.0 (13.09) | 60.1 (16.52)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 3 | 3 | 1 | 11
  Male | 2 | 2 | 3 | 1 | 6 | 2 | 16
  Unknown | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 4 | 1 | 3 | 0 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 4 | 3 | 0 | 3 | 5 | 3 | 18
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 3 | 4 | 4 | 9 | 4 | 28

OUTCOME MEASURES:

1. Primary Outcome: Brain Flortaucipir Uptake
Description: Brain imaging of tau in healthy volunteers and subjects with cognitive impairment. Standard uptake value ratios (SUVr), normalized to the entire cerebellum. A global cortical average volume of interest (VOI) is the average SUVr of the occipital cortex, parietal cortex, and temporal cortex. For SUVr, a value of 1 signifies no flortaucipir activity above background, values greater than 1 signify increasing flortaucipir activity in the brain.
Time Frame: 80-100 minutes postdose
Population: Includes quantitative flortaucipir PET scan results from subjects with a flortaucipir scan in the present study (n=15), plus subjects consented in the MRI/Amyloid extension cohort who provided valid flortaucipir PET scans (n=3 AD, n=2 MCI, n=1 OCN) and received MRI in the present study permitting quantitative analysis per protocol.
Measure: Mean (Standard Deviation); unit: standardized uptake value ratio (SUVr)
Arm/Group | Brain PET Scan (AD Subjects) | Brain PET (MCI Subjects) | Brain PET (YCN Subjects) | Brain PET (OCN Subjects)
Number analyzed (Participants) | 7 | 5 | 4 | 5
standardized uptake value ratio (SUVr) | 1.780 (0.857) | 1.317 (0.161) | 1.128 (0.047) | 1.107 (0.175)

2. Primary Outcome: Flortaucipir Whole Body Effective Dose
Description: Radiation dose estimates measured in millisieverts per megabecquerel (mSv/MBq) for the whole body obtained from Organ Level Internal Dose Assessment/Exponential Modeling (OLINDA/EXM) radiation dosimetry code. Results calculated using 73.7-kg man model.
Time Frame: injection to 6 hours postdose
Population: Includes only subjects from the whole body PET scan group (n=9)
Measure: Mean (Standard Deviation); unit: mSv/MBq
Arm/Group | Whole Body Flortaucipir PET Scan
Number analyzed (Participants) | 9
mSv/MBq | 0.0241 (0.00160)

3. Secondary Outcome: Flortaucipir PET Correlations With Cognitive Assessments (Mini-mental State Exam)
Description: Spearman's correlations between flortaucipir SUVr and cognitive function as measured on the Mini-Mental State Examination (MMSE). MMSE is a 30-point questionnaire that is used to measure cognitive impairment. 0 is the lowest score and 30 is the highest score, indicating normal cognitive function. Lower MMSE scores indicate worsening cognitive function. For this analysis, negative correlation values indicate that higher flortaucipir uptake is associated with decreasing cognitive function and positive correlation values indicate that lower flortaucipir uptake is associated with better cognitive function. 95% confidence interval uses a Fisher's z transformation.
Time Frame: at baseline
Population: Includes quantitative flortaucipir brain PET scan results from subjects with a flortaucipir scan in the present study (n=15), plus subjects consented in the MRI/Amyloid extension cohort who provided valid flortaucipir PET scans from a previous study (n=6) and received MRI in the present study permitting quantitation per protocol.
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Groups:
- All Subjects/Brain PET: Includes all AD, MCI, YCN, and OCN subjects enrolled in the study with flortaucipir Brain PET scans
Arm/Group | All Subjects/Brain PET
Number analyzed (Participants) | 21
correlation coefficient | -0.404 [-0.706 to 0.044]

4. Secondary Outcome: Flortaucipir PET Correlations With Cognitive Assessments Cognitive Assessments (Digit Symbol Substitution Test)
Description: Spearman's correlations between flortaucipir SUVr and cognitive function as measured on Digit Symbol Substitution Test (DSST). The DSST is sensitive to the presence of cognitive dysfunction as well as to change in cognitive function. Scores range from 0 to 133. Lower DSST scores indicate worsening cognitive function. For this analysis, negative correlation values indicate that higher flortaucipir uptake is associated with decreasing cognitive function and positive correlation values indicate that lower flortaucipir uptake is associated with better cognitive function. 95% confidence interval uses a Fisher's z transformation.
Time Frame: at baseline
Population: Includes quantitative flortaucipir PET scan results from subjects with a flortaucipir scan in the present study (n=15), plus subjects consented in the MRI/Amyloid extension cohort who provided valid flortaucipir PET scans from a previous study n=6) and received MRI in the present study permitting quantitation per protocol.
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | All Subjects/Brain PET
Number analyzed (Participants) | 21
correlation coefficient | -0.273 [-0.744 to 0.403]

5. Secondary Outcome: Flortaucipir PET Correlations With Cognitive Assessments Cognitive Assessments (Alzheimer's Disease Assessment Scale)
Description: Spearman's correlations between flortaucipir SUVr and cognitive function as measured on a Modified Alzheimer's Disease Assessment Scale (ADAS)-Cognitive subscale (including orientation, verbal memory, language, and praxis, minus the spoken language assessment). Scores on the modified scale can range from 0 to 65. Higher scores indicate worsening cognitive function. For this analysis, positive correlation values indicate that higher flortaucipir uptake is associated with decreasing cognitive function and negative correlation values indicate that lower flortaucipir uptake is associated with better cognitive function. 95% confidence interval uses a Fisher's z transformation.
Time Frame: at baseline
Population: Includes quantitative flortaucipir PET scan results from subjects with a flortaucipir scan in the present study (n=15), plus subjects consented in the MRI/Amyloid extension cohort who provided valid flortaucipir PET scans from a previous study (n=6) and received MRI in the present study permitting quantitation per protocol.
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | All Subjects/Brain PET
Number analyzed (Participants) | 21
correlation coefficient | 0.220 [-0.447 to 0.719]

6. Post Hoc Outcome: Flortaucipir Whole Body Effective Dose With Urine Radioactivity
Description: Radiation dose estimates measured in millisieverts per megabecquerel (mSv/MBq) for the whole body obtained from Organ Level Internal Dose Assessment/Exponential Modeling (OLINDA/EXM) radiation dosimetry code. Results calculated using 73.7-kg man model and accounting for total integrated radioactivity excreted in the urine collected in Study A15 (NCT02336360)
Time Frame: injection to 6 hours postdose
Population: Includes only subjects from the whole body PET scan group (n=9)
Measure: Mean (Standard Deviation); unit: mSv/MBq
Arm/Group | Whole Body Flortaucipir PET Scan
Number analyzed (Participants) | 9
mSv/MBq | 0.0235 (0.0016)

ADVERSE EVENTS:
Time Frame: End of study for AE reporting was 48 hours after the last study drug administration.
Description: Adverse Events were defined as occurring or worsening after injection of dose, within 48 hours post injection of florbetapir or flortaucipir. AEs occurring after study drug administration, but outside that window were not recorded in the database, unless considered attributable to study drug injection. MRI/Amyloid extension cohort n=4 represents only those subjects receiving florbetapir PET scans.
Groups:
- MRI and Amyloid Extension Cohort: Magnetic resonance imaging (MRI) scans and amyloid scans for subjects previously participating in Study T807000
Arm/Group | Brain PET Scan (AD Subjects) | Brain PET (MCI Subjects) | Brain PET (YCN Subjects) | Brain PET (OCN Subjects) | Whole Body PET Scan | MRI and Amyloid Extension Cohort
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/4 | 0/4 | 0/9 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/4 | 0/4 | 0/9 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 1/4 | 0/4 | 3/9 | 0/4
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brain PET Scan (AD Subjects) (N=4) | Brain PET (MCI Subjects) (N=3) | Brain PET (YCN Subjects) (N=4) | Brain PET (OCN Subjects) (N=4) | Whole Body PET Scan (N=9) | MRI and Amyloid Extension Cohort (N=4)
headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less